CLINICAL TRIAL: NCT00305032
Title: Effect of Endoscopic Gastric Balloon Insertion on Obstructive Sleep Apnea in Patients With Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, To Kin Wang, Doctor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2005.399
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Morbid Obesity; Obstructive Sleep Apnea
MeSH Terms: conditions — Obesity, Morbid; Sleep Apnea, Obstructive | interventions — Gastric Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: gastric balloon insertion

INTERVENTIONS:
Procedure: gastric balloon insertion — patient would be offered endoscopic gastric balloon insertion
  Other Names: gastric balloon

SUMMARY:
To investigate the effect of weight loss by gastric balloon insertion on parameters of obstructive sleep apnea.

DETAILED DESCRIPTION:
Most of the patients with obstructive sleep apnea (OSA) are obese. It has been noted that significant weight loss could improve the severity of sleep apnea. Significant weight loss is difficult to achieve especially in morbidly obese patients. Endoscopic gastric balloon insertion is minimally invasive procedure is employed by surgeon for weight reduction for morbidly obese patients. This study would assess the parameters of sleep which could be affected by weight reduction. If results are positive, this procedure might be considered as treatment for obstructive sleep apnea in morbidly obese patients.

Patient population would be selected from patients who would undergo gastric balloon insertion in the surgical department. There would be no sex or age limit. Patient recruited would have BMI > 35. Consent would be signed for sleep studies. Baseline sleep study, lung function, Epworth Sleepiness Scale (ESS) and quality of life would be assessed in patients who have symptoms suggestive of OSA. If a patient is confirmed to have OSA, a continuous positive airway pressure (CPAP) titration would be offered if the patient is willing to try CPAP. Otherwise patients would be discharged home and wait for balloon insertion. The same assessment would be repeated 3 months and 6 months after the surgical procedure. All sleep studies would be done as in-patient.

Leptin and ghrelin are hormones control satiety, which are also related to the degree of obesity. Blood for plasma leptin and ghrelin would be taken before and 6 months after gastric balloon insertion to assess the relationship of weight reduction by reducing appetite and plasma level of the hormones

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patients with BMI > 30
* confirmed obstructive sleep apnea with RDI > 10/hr
* able to sign consent

Exclusion Criteria:

* patients undergoing weight reduction surgery
* sleep apnea other than obstructive sleep apnea
* untreated endocrine disorder
* patient refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-03; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
effect of gastric balloon on sleep apnea | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: To K Wang, FHKCP, FACCP, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China